CLINICAL TRIAL: NCT04526561
Title: Reconstructions With Back Donor Site Flaps and Validation of Quality of Life Scales
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 254-18
Record Dates: First submitted 2020-08-12; First posted 2020-08-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast reconstruction TDAP (Active Comparator): Breast reconstruction performed with TDAP
  Interventions: Procedure: Thoracodorsal artery perforator flap to breast
- Breast reconstruction latissimus dorsi (Active Comparator): Breast reconstruction performed with latissimus dorsi
  Interventions: Procedure: Latissimus dorsi flap
- Breast reconstruction with DIEP (Active Comparator): Breast reconstruction performed with a deep inferior epigastric artery perforator flap
  Interventions: Procedure: Deep inferior epigastric perforator flap

INTERVENTIONS:
Procedure: Latissimus dorsi flap — Breast reconstruction
  Other Names: LD flap
  Arms: Breast reconstruction latissimus dorsi
Procedure: Thoracodorsal artery perforator flap to breast — Breast reconstruction
  Other Names: TDAP
  Arms: Breast reconstruction TDAP
Procedure: Deep inferior epigastric perforator flap — Breast reconstruction
  Other Names: DIEP flap
  Arms: Breast reconstruction with DIEP

SUMMARY:
The latissimus dorsi flap is the oldest and most used technique for breast reconstruction. Nonetheless, there are few studies evaluation the long-term effect of harvesting one of the muscles of the back. This project has four parts.

1. Validation of scales/instrument for Swedish.
2. Long-term results after reconstruction with latissimus dorsi- a ten year retrospective follow-up.
3. Thoracodorsal artery perforator flap (TDAP) vs latissimus dorsi flap- a randomized controlled trial - breast reconstruction.
4. TDAP vs Limber flap - a randomized controlled trial- reconstruction of axillary hidradenitis suppurativa.

ELIGIBILITY:
Inclusion criteria:

* Patients eligible for breast reconstruction following mastectomy and radiation
* Non-smokers or ex-smokers (>6 weeks)
* BMI < 30

Exclusion Criteria:

* Inability to leave informed consent
* Inability to understand Swedish
* Previous surgery with scaring on back

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological women identifying themselves as cis-women.
Enrollment: 550 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction and breast-related quality of life after breast reconstruction | 10 years
  Breast Q reconstruction.The BREAST-Q has multiple domains, each scored from 0 to 100 (higher scores indicate greater satisfaction or quality of life), there is no overall BREAST-Q score.
Back and shoulder function after breast reconstruction | 10 years
  Breast Q the back and shoulder function scale. The scale is scored from 0 (worst) to 100 (best). Higher scores reflect a better outcome.
Back appearance after breast reconstruction | 10 years
  Breast-Q the back appearance scale.The scale is scored from 0 (worst) to 100 (best). Higher scores reflect a better outcome.
Shoulder function after breast reconstruction | 10 years
  Western Ontario Osteoarthritis of the shoulder index (WOOS) provides scores on four domains: (1) physical symptoms; (2) sport, recreation, and work; (3) lifestyle; and (4) emotions.Each question has a possible score from 0-100 giving a total score up to 1900. The highest or most symptomatic score is 1900 and the best or asymptomatic score is 0.
Abdominal satisfaction after breast reconstruction | 10 years
  Breast Q abdominal satisfaction and abdominal well-being.The scale is scored from 0 (worst) to 100

SECONDARY OUTCOMES:
Complications after breast reconstruction | 2 years
  Measured in patients randomized to TDAP or latissimus dorsi flap.

OTHER OUTCOMES:
Validation of Breast Q: The Back Appearance scale for Swedish | 1 year
  Translation and validation of the instrument for Swedish
Validation of Breast-Q: The back and shoulder function scale for Swedish | 1 year
  Translation and validation of the instrument for Swedish
Normal material for Breast-Q | 5 years
  Measurement of quality of life according to breast-Q in a normative population
Normal material for Breast-Q back appearance scale | 5 years
  Measurement of quality of life according to breast-Q back appaearance scale in a normative population
Normal material for Breast-Q back and shoulder function scale | 5 years
  Measurement of quality of life according to breast-Q back and shoulder function scale in a normative population

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

REFERENCES:
- [Result] Kamya L, Hansson E, Weick L, Hansson E. Validation and reliability testing of the Breast-Q latissimus dorsi questionnaire: cross-cultural adaptation and psychometric properties in a Swedish population. Health Qual Life Outcomes. 2021 Jul 3;19(1):174. doi: 10.1186/s12955-021-01812-x. PMID 34217326